CLINICAL TRIAL: NCT03491787
Title: Ultrasound-guidance for Intraosseous Access Could Provide Benefits for Resuscitation in Out-of-hospital Traumatic Cardiac Arrest: a Field Report During Earthquake on Amatrice (Italy), August 24, 2016
Brief Title: Ultrasound-guidance for Intraosseous Access During Earthquake
Status: Completed | Type: Observational
Sponsor: San Salvatore Hospital of L'Aquila (Other)
Responsible Party: Principal Investigator, Emiliano Petrucci, Medical Doctor of Anesthesia and Intensive Care Unit, San Salvatore Hospital of L'Aquila
Other Study IDs: 05/01/2017, n.12
Record Dates: First submitted 2018-03-28; First posted 2018-04-09 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Arrest Due to Trauma (Disorder)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Ultrasound guidance: The ultrasound guidance was used to establish intraosseous access
  Interventions: Device: Ultrasound guidance
- Not ultrasound guidance: The ultrasound guidance was not used to obtain intraosseous access

INTERVENTIONS:
Device: Ultrasound guidance — The ultrasound guidance was used to obtain intraosseous access
  Groups: Ultrasound guidance

SUMMARY:
The aim of this field report is to describe as the use ultrasound guidance can facilitate the insertion of intraosseous access, during the resuscitation, in the victims of out-of hospital traumatic cardiac arrest

DETAILED DESCRIPTION:
The aim of this field report is to describe as the use ultrasound guidance can facilitate the insertion of intraosseous access, decreasing the time for drug administration and providing some benefits during the resuscitation, in the victims of out-of hospital traumatic cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* traumatic cardiac arrest

Exclusion Criteria:

* non traumatic cardiac arrest
* beheading
* post-mortem hypostasis
* carbonized bodies
* dismembered bodies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People under the rubble, after the earthquake
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-09-26 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Intraosseus access | up to 10 minutes
  The time used to esteblish the intraosseus access

SECONDARY OUTCOMES:
Return of spontaneous circulation | up to 1 hour
  The time to obtain the return of spontaneous circulation